CLINICAL TRIAL: NCT01064661
Title: Physiological Effects of Probiotic Bacteria Lactobacillus Acidophilus NCFM Alone Versus a Combination With Bifidobacterium Lactids - LBi07 in Patients With Mild to Moderate Abdominal Pain/Discomfort and Bloating
Brief Title: Pilot Study Studying Physiological Effects of Probiotic Pills in Patients With Abdominal Pain/Discomfort and Bloating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Danisco (Industry)
Responsible Party: Principal Investigator, Yehuda Ringel, Associate Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 09-0337
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Abdominal Pain; Abdominal Discomfort; Bloating; Functional Bowel Disorders
Keywords: Probiotics; abdominal pain; abdominal discomfort; bloating; Functional Bowel Disorders
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blend probiotic of L-NCFM and B-LBi07 (Active Comparator): Blend probiotic pills of L-NCFM and B-LBi07 BID (2x10^10 cfu total bacteria per day)
  Interventions: Dietary Supplement: Blend probiotic arm of L-NCFM and B-LBi07
- Single probiotic of L-NCFM alone (Active Comparator): Single probiotic pills of L-NCFM alone BID (2x10^10 cfu total bacteria per day)
  Interventions: Dietary Supplement: Single probiotic arm of L-NCFM alone

INTERVENTIONS:
Dietary Supplement: Single probiotic arm of L-NCFM alone — Single probiotic of L-NCFM alone pills BID (2x10^10 cfu total bacteria per day)
  Other Names: Lactobacillus Acidophilus NCFM
  Arms: Single probiotic of L-NCFM alone
Dietary Supplement: Blend probiotic arm of L-NCFM and B-LBi07 — Blend probiotic arm of L-NCFM and B-LBi07 pills BID (2x10^10 cfu total bacteria per day)
  Other Names: Lactobacillus Acidophilus NCFM; Bifidobacterium Lactids - LBi07
  Arms: Blend probiotic of L-NCFM and B-LBi07

SUMMARY:
We are conducting a study to learn if probiotics, which are live bacteria found in food like yogurt and cheese, will improve symptoms of abdominal pain. Individuals participating in this study will take probiotic pills to see if this affects the expression of certain pain receptors in the intestines that relate to pain sensation. Biopsies will be taken from the colon before subjects take the probiotic pills. Subjects will then be given one of two different types of probiotic pills to take for 3-4 weeks. After taking the supplements, more biopsies will be collected to see if any changes have taken places. This study requires one screening visit and two clinic visits to UNC hospital. Subjects will also complete daily diary cards for 2 weeks during the study to record their symptoms and also collect 2 stool samples.

DETAILED DESCRIPTION:
The purpose of this study is to determine if probiotic bacteria, specifically Lactobacillus and Bifidobacterium, have an effect on pain receptors in the colon. Data from animal studies suggest that daily consumption of probiotic bacteria can increase expression of specific receptors in the intestinal mucosa in mice and that these mucosal effects are associated with decrease in intestinal pain sensation. We are interested to see if this is true in humans as well.

Probiotics are live bacteria, which can be found in certain foods like yogurt or cheese prepared with active cultures. The use of probiotics has been shown to be successful in several intestinal disorders, including chronic inflammatory bowel disease (IBD), childhood diarrhea (rotavirus infection), and travelers' diarrhea. This has led to increased interest in their use in patients with symptoms of abdominal pain or discomfort. Although, the data on the use of probiotics in bloating is limited, several reported studies show encouraging results and suggest a symptomatic response and parallel improvement in quality of life.

Probiotics are regarded by the US Food and Drug Administration (FDA) as dietary supplements. They do not require approval by the FDA or any government agency prior to marketing however they are subjected to the FDA jurisdiction regarding their safety, labeling, and health statements. Probiotics can be provided in various forms including food (such as yogurt) or in the format of pills, tablets, caps, and liquids. In this study they will be given in a pill form.

You are being asked to participate in this study because you are currently experiencing abdominal pain or discomfort in your abdomen and you have a functional bowel disorder. In order to determine if these probiotics have an effect, you will be asked to either take a Bifidobacterium probiotic or a blend of Bifidobacterium plus Lactobacillus probiotic. You will be asked to undergo an un-prepped, un-sedated flexible sigmoidoscopy both before your treatment course and after your treatment course. Biopsy samples will be taken during this procedure to analyze certain pain receptor levels, comparing differences between the two treatments of probiotics, and differences in receptors before after treatment. We may use this data for future research in understanding the probiotic function in the gut. We may also perform genetic testing on these specimens in order to look for relationships between genes, the environment, and people's habits or diet, and different diseases. All remaining samples will be stored for-as-yet-unknown tests.

Please note that in order to participate in this study the separate storage consent form is non-optional and must be signed allowing long term storage of stool samples.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent has been signed.
2. The subject is a female.
3. The subject is 18 - 70 years old.
4. Active symptoms of abdominal pain or discomfort. Other functional bowel disorders including IBS, functional abdominal pain, and functional bloating are also allowed. For all functional bowel disorders we will use the definition provided by the Rome III criteria.
5. The subject's abdominal pain is of mild to moderate in severity. Severity of abdominal pain will also be determined using 10 point likert scale.
6. Subjects > 50 years old must have had a screening colonoscopy with a normal report in the past 5 years - per subject report at time of phone screen. Removal of polyps and hemorrhoids are acceptable.

Exclusion Criteria:

1. The subject has inflammation or structural abnormality of the digestive tract [e.g. inflammatory bowel disease (IBD), duodenal ulcer (DU) or gastric ulcer (GU), obstruction, or symptomatic cholelithiasis.
2. The subject has severe abdominal pain symptoms at baseline.
3. The subject has a serious, unstable medical condition, such as lung disease, uncontrolled blood pressure, uncontrolled thyroid function, a physical or medical disability or an advanced medical condition.
4. The subject has insulin-dependent Diabetes Mellitus.
5. The subject had a major psychiatric diagnosis or a suicide attempt within the last two years.
6. The subject has a history of alcohol or substance abuse within two years.
7. The subject has been treated for a malignancy within the last 5 years (except BCC or SCC skin cancer).
8. The subject has been diagnosed with lactase deficiency and this can explain their symptoms (i.e., symptoms resolved or reduced significantly with lactose-free diet.)
9. The subject had previous significant gastric or intestinal surgery (except appendectomy and gall bladder surgery).
10. Subject is pregnant or lactating, or planning to become pregnant. (A urine pregnancy test will be performed on female subjects prior to the flexible sigmoidoscopy procedure. Acceptable forms of birth control include oral contraceptives, double barrier method, and IUD cover and must be practiced from the time of enrollment until the time of release from the study.)
11. The subject is predisposed to infection (i.e. their immune system is compromised, they have rheumatic heart disease, an artificial valve, history of bacterial endocarditis, or an active bacterial disease)
12. The subject received antibiotic treatment or was intentionally consuming probiotic supplementation on a daily basis during the last 4 weeks. If a subject uses antibiotics or probiotics, a 4 weeks washout period is required prior to enrollment.
13. The subject has taken medication for pain relief or anti-inflammatory medications (e.g., aspirin, NSAID, or steroids) in the last 10 days. If a subject uses pain medication or anti-inflammatory medications, a 10 days washout period is required prior to enrollment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Investigate/compare the effect of the probiotic bacteria L-NCFM alone or in combination with B-LBi07 on expression of intestinal mucosal receptors involved in transmission of nociceptive information. | 21-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ringel, MD, Principal Investigator — UNC Dept. Gastroenterology and Hepatology

REFERENCES:
- [Background] Rousseaux C, Thuru X, Gelot A, Barnich N, Neut C, Dubuquoy L, Dubuquoy C, Merour E, Geboes K, Chamaillard M, Ouwehand A, Leyer G, Carcano D, Colombel JF, Ardid D, Desreumaux P. Lactobacillus acidophilus modulates intestinal pain and induces opioid and cannabinoid receptors. Nat Med. 2007 Jan;13(1):35-7. doi: 10.1038/nm1521. Epub 2006 Dec 10. PMID 17159985
- [Derived] Ringel-Kulka T, Goldsmith JR, Carroll IM, Barros SP, Palsson O, Jobin C, Ringel Y. Lactobacillus acidophilus NCFM affects colonic mucosal opioid receptor expression in patients with functional abdominal pain - a randomised clinical study. Aliment Pharmacol Ther. 2014 Jul;40(2):200-7. doi: 10.1111/apt.12800. Epub 2014 May 22. PMID 24853043